CLINICAL TRIAL: NCT04627376
Title: Effectiveness of a Multimodal Education and Support Program for the Prevention of Cancer Related Cachexia for Patients and Their Family Caregiver
Brief Title: Multimodal Program for Cancer Related Cachexia Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: German Oncology Center, Cyprus (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Associate Professor Oncology and Palliative Care, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CC-SPCC-1
Record Dates: First submitted 2020-10-27; First posted 2020-11-13 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Neoplasms; Cancer; Cachexia; Malnutrition; Educational Problems
Keywords: cachexia; prevention; management; malnutrition
MeSH Terms: conditions — Neoplasms; Cachexia; Malnutrition | interventions — MME

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 12-weeks multimodal program includes: 4 meetings (with cancer nurse and clinical dietician). In this 4 meetings (about 30 minutes) they will have blood tests (CRP, Albumin levels), body composition measurements, questionnaires.
- Intervention (Experimental): 12-weeks multimodal program includes: 4 meetings (with cancer nurse and clinical dietician). In this 4 meetings (about 30 minutes) they will have blood tests (CRP, Albumin levels), body composition measurements, questionnaires, education on their diet and symptom management related to anti cancer treatment.
  Interventions: Other: Multimodal education and support program for cancer related cachexia prevention

INTERVENTIONS:
Other: Multimodal education and support program for cancer related cachexia prevention — 12-weeks multimodal program includes: 4 meetings (with cancer nurse and clinical dietician). In this 4 meetings (about 30 minutes) they will have blood tests (CRP, Albumin levels), body composition measurements, questionnaires, education on their diet and symptom management related to anti cancer treatment.
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate the effectiveness of a multifactorial education and support program for the prevention of cancer-related cachexia syndrome, for patients and their family caregivers during anti-cancer treatment.

DETAILED DESCRIPTION:
After being informed about the study and the need to nominate a family caregiver, all patients and their family caregiver giving written informed consent, they will undergo a 12-weeks multimodal program. Randomly they will divided into two groups (intervention and control). This 12-weeks multimodal program includes 4 meetings (with cancer nurse and clinical dietician). In this 4 meetings (about 30 minutes) they will have blood tests (CRP, Albumin levels), body composition measurements, questionnaires, education on their diet and symptom management.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Participants must be diagnosed with solid tumour (stomach, colorectal, pancreas, breast, lung)
3. Participants needing chemotherapy/immunotherapy/hormone therapy/target therapy
4. Participants must be normal or pre cachectic as defined by the guidelines
5. Read and understand Greek or English

Exclusion Criteria:

1. Haematologic tumors
2. Parenteral Nutrition
3. ECOG Performance status >2 or Karnofsky Performance Status <60%
4. Participant who can not introduce a family caregiver
5. Participants in cachexia or refractory cachexia stage as defined by the guidelines below:

   * >5% weight loss over the past 6 months (in absence of simple starvation); OR
   * BMI <20 and any degree of weight loss >2%; OR
   * Appendicular skeletal muscle index consistent with sarcopenia (whole body fat-free mass index without bone determined by bioelectrical impedance (men <14.6 kg/m²; women <11.4 kg/m²) and weight loss >2%
6. Patients who use complementary therapies (ex-acupuncture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-cachexia stage against cachexia criteria at 12 weeks | Baseline and week 4, week 8, week 12
  To assess the patient's baseline cancer cachexia stage with weight (weight loss <5% in previous three months, kg), height (cm) and BMI (BMI > 20) measurements.

SECONDARY OUTCOMES:
Change from baseline in inflammation based on the CRP test at 12 weeks | Baseline and week 4, week 8, week 12
  Blood test for C-reactive protein (mg/L). CRP level greater than 10 mg/L is a sign of active inflammation.
Change from baseline in edema according to albumin levels from baseline at 12 weeks | Baseline and week 4, week 8, week 12
  Blood test for Albumin Levels. normal ranges >35g/L
Change from baseline of patient's Quality of life on the FAACT questionnaire (score) at 12 weeks | Baseline and week 12
  Participants will fill the questionnaire at baseline and at week 12 to compare the score of FAACT.
  The FAACT questionnaire is validated, self-reported instrument (28-item) assessing the quality of life of cancer patients with any tumour type. Possible scores range from 0 (lower quality of life) to 112 (better quality of life).
  Change = Week 12 - Baseline
Change from baseline (week 4) of family caregiver's Quality of life on the CarGOQoL questionnaire (score) at 12 weeks | Week 4 and week 12
  Participants will fill the questionnaire at week 4 and at week 12 to compare the score of CarGOQoL.
  The CarGOQoL questionnaire is validated, self-reported instrument (29 items investigating 10 domains) assessing the quality of life of family caregivers. Possible scores range from 0 (lower quality of life) to 100 (better quality of life).
  Change = Week 12 - Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Study Director — Cyprus University of Technology Department of Nursing
Locations (1):
- German Oncology Centre, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No